CLINICAL TRIAL: NCT06808880
Title: EXpanding Prenatal Cell Free DNA Screening Across moNogenic Disorders (EXPAND)
Acronym: EXPAND
Status: Recruiting | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 23-075-WH
Record Dates: First submitted 2025-01-21; First posted 2025-02-05 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-02

CONDITIONS: Single Gene NIPT
Keywords: single gene NIPT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A whole blood sample will be collected from the pregnant participant. If prenatal diagnostic testing results or clinical testing results are not available or are uninformative for the single-gene disorder of interest, a newborn cheek swab will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Increased Risk for Single Gene Disorder
  Interventions: Device: Single-gene Noninvasive Prenatal Testing (sgNIPT)

INTERVENTIONS:
Device: Single-gene Noninvasive Prenatal Testing (sgNIPT) — Natera sgNIPT is intended for use in pregnant people whose 'fetus/ fetuses are identified as at increased risk for a single gene disorder when there is no reproductive partner (paternal) screening available or when there is positive reproductive partner screening, but prenatal diagnostic testing is not an option or when there is concern for a single-gene disorder in the fetus/ fetuses irrespective of carrier status (e.g., based on fetal ultrasound findings).

SUMMARY:
The purpose of this research is to develop and validate a single gene Non-Invasive Prenatal Test. The development of this investigational single-gene noninvasive prenatal testing (sgNIPT) for conditions such as cystic fibrosis (CF), spinal muscular atrophy (SMA), Sickle cell disease, alpha thalassemia (a-thalassemia) and beta thalassemia (b-thalassemia) could provide information about the possibility that a child will be born with a serious health condition, in some cases in the absence of reproductive partner screening.

In order to develop a test for this purpose, investigators will collect blood samples and medical information from pregnant women who have pregnancies at higher risk for single gene disorders, such as those who are carriers for these conditions or affected by these conditions themselves, medical data from their reproductive partners in some cases, and either genetic testing results or a cheek swab sample from the newborn(s).

DETAILED DESCRIPTION:
Natera sgNIPT is intended for use in pregnant people whose fetus/ fetuses are identified as at increased risk for a single gene disorder, such as one of the disorders below, when there is no reproductive partner (paternal) screening available or when there is positive reproductive partner screening, but prenatal diagnostic testing is not an option or when there is concern for a single-gene disorder in the fetus/ fetuses irrespective of carrier status (e.g., based on fetal ultrasound findings). Disorders include:

CF (CFTR) SMA (SMN1) Alpha-thalassemia (HBA1/HBA2) Beta-hemoglobinopathies including sickle cell disease (HBB)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older at the time of informed consent
2. Maternal participant: Pregnant and blood draw at ≥ 9 weeks gestational age (GA)
3. Maternal participant is positive for a single-gene disorder and/or there are prenatal ultrasound findings suggestive for a fetal single-gene disorder, including but not limited to the genes listed in the primary and secondary objectives
4. Meet the criteria for one of the following:

   * Both maternal and reproductive partner (paternal) status are positive for the same single-gene disorder OR
   * A commercially available single-gene NIPT has been performed as part of clinical care and is reported as increased risk for an affected fetus/fetuses OR Maternal status is positive for one or more single-gene disorders and reproductive partner status is unknown OR
   * Prenatal ultrasound findings are suggestive of a fetal single-gene disorder (autosomal dominant, autosomal recessive, or X-linked condition) and enrollment is approved by the medical monitor.
5. Willing to permit release of neonatal health information and the performance of a newborn cheek swab within 6 months following delivery
6. Willing to sign informed consent and comply with study procedures

Exclusion Criteria:

1. Reproductive partner found to not be positive for the same autosomal recessive genetic disorder as the pregnant maternal carrier, or vice versa
2. Surrogate gestation or egg donor pregnancy
3. Negative preimplantation genetic testing for the single-gene disorder identified in one or both parents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Natera sgNIPT is intended for use in pregnant people whose fetus/ fetuses are identified as at increased risk for a single gene disorder when there is no reproductive partner (paternal) screening available or when there is positive reproductive partner screening but prenatal diagnostic testing is not an option or when there is a concern for single-gene disorder in the fetus/ fetuses irrespective of carrier status (e.g., based on fetal ultrasound findings).
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Performance of sgNIPT assay in the detection of primary four autosomal recessive disorders | Following the development of the sgNIPT assay, approximately 2 years after the launch of the study
  The sgNIPT assay call, high risk or low risk; will be compared to the genetic outcome of the fetus/ fetuses Affected; or Not Affected; as determined by prenatal genetic testing, post-natal genetic testing or genetic testing performed on the newborn cheek swab sample. Sensitivity, PPV, NPV, and no call rates will be assessed.

SECONDARY OUTCOMES:
Performance of sgNIPT assay in the detection of single gene disorders other than the primary four | Following the development of the primary disorder assay, approximately 2.5 years after the launch of the study
  The sgNIPT assay call, high risk or low risk; will be compared to the genetic outcome of the fetus/ fetuses Affected; or Not Affected; as determined by prenatal genetic testing, post-natal genetic testing or genetic testing performed on the newborn cheek swab sample. Sensitivity and PPV pooled across single gene disorders other than the four primary disorders

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Valley Perinatal, Glendale, Arizona
  - Cedars Sinai Prenatal Diagnosis Center, Los Angeles, California
  - Center for Fetal Medicine and Womens Ultrasound, Los Angeles, California
  - Natera Inc, San Carlos, California
  - University of California San Francisco, San Francisco, California
  - Orlando Health Inc. (Winnie Palmer Hsopital), Orlando, Florida
  - UMMC WH Univerity Center For Fetal Medicine, Jackson, Mississippi
  - Capital Health, Lawrenceville, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - NYU Langone Hospital, Garden City, New York
  - Northwell (Northshore/LIJ), New Hyde Park, New York
  - NYU Langone, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Austin Maternal Fetal Medicine/St. Davids Healthcare, Austin, Texas
  - University of Texas Medical Branch (UTMB), Galveston, Texas
  - PEDIATRIX Medical Services, Inc. Master + Houston, Stafford, Texas

IPD SHARING:
Plan to Share IPD: No
This study is for the development of a proprietary product, therefore the individual data will not be shared.

REFERENCES:
- See also: Page for potential participants to learn about the study and express interest in participating — https://www.natera.com/info/expand-study/